CLINICAL TRIAL: NCT05749627
Title: A Clinical Study of Personalized Tumor Neoantigen Peptide Vaccine/neoantigen-based Dendritic Cells in the Treatment of Advanced Malignant Solid Tumors
Brief Title: Using Neoantigen Peptide Vaccine/neoantigen-based DC to Treat Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Collaborators: Shanghai Dengding BioAI Co. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2021-087
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Neoantigen Peptide Vaccine; Neoantigen-based Dendritic Cells; Therapeutic immune preparation; Advanced Malignant Solid Tumors; Progression-free Survival; Overall Survival; Overall Response Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoantigen peptide vaccine/neoantigen-based DC treatment (Experimental): Patients assigned to the neoantigen peptide vaccine/neoantigen-based DC treatment group will receive 5-6 subcutaneous injections of neoantigen peptide vaccine or neoantigen-based DC immune preparation within a 14-week treatment period.
  Interventions: Drug: Neoantigen peptide vaccine; Drug: Neoantigen-based DC immune preparation

INTERVENTIONS:
Drug: Neoantigen peptide vaccine — Personalized tumor neoantigen peptide vaccine
Drug: Neoantigen-based DC immune preparation — Personalized tumor neoantigen DC therapeutic immune preparation

SUMMARY:
In this study, the investigators provide a personalized tumor neoantigen peptide vaccine/neoantigen-based DC treatment to patients with advanced malignant solid tumors. The investigators observe the post-treatment tumor burden status, the immune response induced by immune preparations, and the prolongation of patient survival time, aiming to evaluate the effectiveness and safety of the neoantigen-based DC treatment.

DETAILED DESCRIPTION:
This study is conducted in accordance with the Declaration of Helsinki and the guidelines of the Consolidated Standards of Reporting Trials.

20 patients with primary or metastatic melanoma, gastrointestinal tumor, breast cancer, cervical cancer, pancreatic cancer, lung cancer, or other malignant tumors will be recruited in this study. With doctor's assessment, a personalized tumor neoantigen peptide vaccine or neoantigen-based DC treatment plan will be designed for each participant：

1. Collecting venous blood samples;
2. Blood PBMC exome sequencing;
3. RNA transcriptome sequencing;
4. Classifying HLA alleles;
5. Performing bioinformatics analysis, finding meaningful mutations and about 10 neoantigen sequences for each patient;
6. Synthesizing peptide neoantigens;
7. Preparation of the personalized tumor neoantigen peptide vaccine or generating the personalized tumor neoantigen DC therapeutic immune preparation.

Participants will receive 5-6 subcutaneous injections of the vaccine or DC preparation within a treatment period of 14 weeks. After treatment, participants will have 3 follow-up visits during 9-months. Venous blood collection, physical examination, ECOG Performance Status Scale assessment, CT/MRI scan, X-ray examination, laboratory examination, and other necessary examinations are required at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* With inoperable advanced malignant solid tumors, including melanoma, gastrointestinal tumor, breast cancer, pancreatic cancer, cervical cancer, lung cancer, etc.
* Failed in standard treatment or voluntarily give up other treatment, and been longer than 2 weeks from the end of the last anti-tumor treatment
* Had disease progression prior to treatment
* Expected survival ≥ 3 months
* ECOG performance status of 0, 1, or 2
* With a negative pregnancy test for females of childbearing age
* Able to take effective contraceptive measures and ensure that there is no birth plan within half a year of the study
* Not positive for HIV, HBV, HCV, or TP
* ALT/AST ≤ 2.5 times the upper limit of normal
* ALP ≤ 2.5 times the upper limit of normal
* Serum creatinine ≤1.6 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* In the absence of granulocyte colony-stimulating factor support, proportion of lymphocytes > 20%, absolute neutrophil count ≥ 1x10^9/L, white blood cell count ≥ 3x10^9/L, platelet count ≥ 100×10^9/L, hemoglobin > 8.0 g/dL, CD4+ cell count > 200/μL
* With normal coagulation test and ECG
* Able to understand and willing to sign a written informed consent form

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with brain metastases
* Had immunosuppressant therapy within 1 month or received other immunotherapy within 3 months
* Participated in other clinical study within 30 days
* With severe allergies or histories of severe allergy
* With splenectomy
* With primary or secondary immunodeficiency diseases or autoimmune diseases (including systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, psoriasis, uncontrolled asthma, etc.)
* Had oral, intramuscular, or intravenous corticosteroids within 1 month. However, inhaled corticosteroids are allowed to treat respiratory insufficiency (such as chronic obstructive pulmonary disease), as well as topical steroids
* With uncontrollable epilepsy, central nervous system disorder, or neurological disease with loss of cognitive ability
* With a history of chronic alcohol or drug abuse within 6 months
* With unstable systemic diseases (including active infection, liver cirrhosis, chronic renal failure, severe chronic pulmonary disease, unstable hypertension, unstable angina, congestive heart failure, myocardial infarction within 1 year, etc.)
* With a history of other malignant tumors in the past 5 years (excluding those who have been clinically cured, and squamous cell carcinoma or skin basal cell carcinoma)
* Those the researcher believed inappropriate to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 9 months after treatment
  Progression-free survival (PFS) is the time from the inoculation of the individualized neoantigen immune preparation to disease progression or death from various causes for all patients. Tumor assessment is performed according to the RECIST1.1 standard. The analysis of this indicator includes results of tumor assessments performed during the treatment period and the follow-up period. If a patient has several indicators that can be judged as disease progression (PD), the indicator that appears first will be used for PFS analysis. Relapse, new tumors, or death are considered to have reached the end of the study. For patients who had not experienced disease progression at the end of the study, the last time the patient had no disease progression was used as censoring data.
Overall response rate | 1 week after treatment
  Overall response rate is the proportion of patients whose tumor shrinkage reaches a certain amount and remains for a certain period of time, including complete response (CR) and partial response (PR) cases. Response Evaluation Criteria in Solid Tumors (RECIST 1.1) was used to evaluate the objective response of tumors. Subjects must have measurable tumor lesions at baseline, and the efficacy evaluation is divided into complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD).
Tumor makers | 9 months after treatment
  CEA，CA19-9，CA125

SECONDARY OUTCOMES:
Overall survival | 9 months after treatment
  Overall survival is the time from inoculation of the individualized neoantigen immune preparation to death due to various causes for all patients.
Disease control rate | 1 week after treatment
  Disease control rate is the percentage of patients who have a complete response (CR), partial response (PR), and stable disease (SD) to the treatment.
Tumor imaging | 9 months after treatment
  CT/MRI scan, X-ray examination etc.
Peripheral blood cytokines | 9 months after treatment
  Changes in peripheral blood cytokines after treatment, including IFN-γ, TNF, IL-2, etc.
ECOG | 9 months after treatment
  Eastern Cooperative Oncology Group (ECOG) Performance Status Scale. This scale describes patients' level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Researchers worldwide consider the ECOG Performance Status Scale when planning cancer clinical trials to study new treatments. There are 6 grades in ECOG, the minimum value is 0 and the maximum value is 5, while a higher score indicates a worse condition.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided